CLINICAL TRIAL: NCT02250703
Title: Comparing Intranasal Dexmedetomidine With Oral Midazolam as Premedication for Older Children Undergoing General Anesthesia for Dental Rehabilitation
Brief Title: Intranasal Dexmedetomidine Premedication in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Madhankumar Sathyamoorthy, Assistant Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014-0131
Record Dates: First submitted 2014-09-05; First posted 2014-09-26 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Preoperative Sedation
Keywords: Premedication
MeSH Terms: interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam (Active Comparator): In M group, patients will be given oral midazolam 0.5mg/kg upto maximum dose of 15mg (5mg/ml parenteral preparation) mixed with flavored syrup as premedication
  Interventions: Drug: Midazolam
- Dexmedetomidine (Experimental): In D group, patients will be given intranasal dexmedetomidine 2mcg/kg upto maximum dose of 100mcg prepared from 100mcg/ml parenteral preparation (Hospira R) . The drug will be administered using a intranasal mucosal administration device (LMA MAD NasalTM).
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Midazolam — oral midazolam 0.5mg/kg upto maximum dose of 15mg
  Arms: Midazolam
Drug: Dexmedetomidine — intranasal dexmedetomidine 2mcg/kg upto maximum dose of 100mcg
  Arms: Dexmedetomidine

SUMMARY:
BACKGROUND INFORMATION AND RATIONALE

Pediatric patients scheduled for dental procedures under general anesthesia can have significant anxiety before the procedure. They are commonly pre medicated to minimize distress and to facilitate a smooth induction of anesthesia. Oral Midazolam at 0.5mg/kg dose is more widely used for this purpose . However the commonly used maximum dose is up to 15mg. It also has many limitations such as paradoxical reaction, increased incidence of emergence delirium and negative postoperative behavior changes . Intranasal dexmedetomidine has been used an effective and safe alternative premedication to oral midazolam in children. At a dose of 2micrograms/kg, intranasal dexmedetomidine as premedication resulted in excellent sedation in children aged 5-8yrs with no adverse hemodynamic effects. It has other advantages such as providing analgesia and facilitating smooth emergence from anesthesia.

The goal of this study is to find out if intranasal dexmedetomidine is a superior alternative as premedication to oral midazolam in children weighing more than 20kg undergoing general anesthesia for dental rehabilitation.

DETAILED DESCRIPTION:
After Institutional Review Board (IRB) approval and written informed consent from patients' parents or legally authorized representative, 80 children older than 5yrs and weighing more than 20kg, ASA physical status 1 or 2, scheduled for elective dental rehabilitation with general anesthesia will be enrolled in this prospective randomized double blinded study.

Exclusion criteria include known allergy or hypersensitivity to midazolam or dexmedetomidine, uncorrected congenital heart disease or history of cardiac arrhythmia, children at risk for airway obstruction (OSA or cranio facial syndrome) and pregnant minors Patients will be randomly assigned to one of two groups M (midazolam) or D (dexmedetomidine) using computer-generated numbers in sealed envelopes.

All the patients will be brought to their pre-op room and premedicated at least 30 min before induction of anesthesia.

In M group, patients will be given oral midazolam 0.5mg/kg upto maximum dose of 15mg (5mg/ml parenteral preparation) mixed with flavored syrup.

In D group, patients will be given intranasal dexmedetomidine 2mcg/kg upto maximum dose of 100mcg prepared from 100mcg/ml parenteral preparation (Hospira R). The drug will be administered using a intranasal mucosal administration device (LMA MAD NasalTM). Atomized nasal medications offer rapid absorption across mucosal membranes to the blood stream avoiding first-pass metabolism.

Parents will be present in the room during premedication. The Anesthesia personnel involved in the care of the patient (MD or CRNA) will prepare and administer all study drugs. All patients will be continuously monitored in the holding area with pulse oximetry and blood pressure monitor. HR, SPO2 and BP will be recorded every 15min after administration of premedication until transfer to the OR. Emergency medications including atropine and epinephrine will be immediately available in the pre-op holding area. Oral midazolam has been used with very little effect on hemodynamic parameters. Although intranasal dexmedetomidine can decrease HR and BP, it has been used at the dose of 2mcg/kg without any adverse hemodynamic effect . Any intervention needed to treat drop in HR (<50) and BP (sys BP <60) after the drug administration will be recorded.

Behavior of the children at the time of premedication will be documented ( easy or difficult). Any unwanted effects during administration such as spitting or vomiting of oral drug and pain or irritation from nasal administration will be documented.

The dental resident blinded to study drug administration will do the pre-operative sedation status and acceptance of mask induction.

Sedation status will be assessed using University of Michigan sedation scale (UMSS)on separation from parents and at induction after moving to the OR table. Acceptance of mask induction will be documented on a 4-point scale.

Standard ASA monitors will be applied before induction of anesthesia. All patients will undergo mask induction with O2/N2O/Sevo. An intravenous line will be inserted and secured. Both nostrils will be prepped nasal drops and tips of tracheal tubes covered with red rubber to minimize bleeding. Nasal intubation will be performed with direct laryngoscopy and McGill's forceps. Appropriate size cuffed tracheal tubes will be inserted and secured after additional IV medications with propofol 2-3mg/kg and fentanyl 1-2mcg/kg. Anesthesia will be maintained with O2/Sevo, IV morphine 0.05 to 0.1mg/kg and IV toradol 0.5mg/kg (if there is no allergy or contraindication to morphine or toradol) After the completion of procedure, patients will be extubated in the operating room and brought to recovery room and allowed to wake up slowly in the recovery position.

PACU nurses will evaluate Behavior at awakening using four-point wake up score (9,20). Patients will also be asked if they remember mask induction (yes or no) when they are ready for discharge. Incidence of nausea, vomiting, shivering will be documented in PACU. Time spent in phase 1 recovery room will also be recorded .

ELIGIBILITY:
Inclusion Criteria:

* Children older than 5yrs and weighing more than 20kg , who are scheduled for ambulatory dental rehabilitation at Batson operating rooms.
* ASA classification 1 or 2

Exclusion Criteria

* Known allergy to midazolam, dexmedetomidine,morphine, fentanyl, sevoflurane and propofol.
* uncorrected congenital heart disease or history of cardiac arrhythmia,
* children at risk for airway obstruction (OSA or cranio facial syndrome),
* pregnant minors

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhankumar Sathyamoorthy, MBBS, MS, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- Children's of Mississippi/University of Mississipi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Background] Kain ZN, Mayes LC, Bell C, Weisman S, Hofstadter MB, Rimar S. Premedication in the United States: a status report. Anesth Analg. 1997 Feb;84(2):427-32. doi: 10.1097/00000539-199702000-00035. PMID 9024042
- [Background] Lonnqvist PA, Habre W. Midazolam as premedication: is the emperor naked or just half-dressed? Paediatr Anaesth. 2005 Apr;15(4):263-5. doi: 10.1111/j.1460-9592.2005.01600.x. No abstract available. PMID 15787915
- [Background] Kanegaye JT, Favela JL, Acosta M, Bank DE. High-dose rectal midazolam for pediatric procedures: a randomized trial of sedative efficacy and agitation. Pediatr Emerg Care. 2003 Oct;19(5):329-36. doi: 10.1097/01.pec.0000092578.40174.85. PMID 14578832
- [Background] McGraw T, Kendrick A. Oral midazolam premedication and postoperative behaviour in children. Paediatr Anaesth. 1998;8(2):117-21. doi: 10.1046/j.1460-9592.1998.00724.x. PMID 9549736
- [Result] Kain ZN, Caldwell-Andrews AA, Krivutza DM, Weinberg ME, Wang SM, Gaal D. Trends in the practice of parental presence during induction of anesthesia and the use of preoperative sedative premedication in the United States, 1995-2002: results of a follow-up national survey. Anesth Analg. 2004 May;98(5):1252-9, table of contents. doi: 10.1213/01.ane.0000111183.38618.d8. PMID 15105196
- [Result] Yuen VM, Hui TW, Irwin MG, Yuen MK. A comparison of intranasal dexmedetomidine and oral midazolam for premedication in pediatric anesthesia: a double-blinded randomized controlled trial. Anesth Analg. 2008 Jun;106(6):1715-21. doi: 10.1213/ane.0b013e31816c8929. PMID 18499600
- [Result] Akin A, Bayram A, Esmaoglu A, Tosun Z, Aksu R, Altuntas R, Boyaci A. Dexmedetomidine vs midazolam for premedication of pediatric patients undergoing anesthesia. Paediatr Anaesth. 2012 Sep;22(9):871-6. doi: 10.1111/j.1460-9592.2012.03802.x. Epub 2012 Jan 23. PMID 22268591
- [Result] Sheta SA, Al-Sarheed MA, Abdelhalim AA. Intranasal dexmedetomidine vs midazolam for premedication in children undergoing complete dental rehabilitation: a double-blinded randomized controlled trial. Paediatr Anaesth. 2014 Feb;24(2):181-9. doi: 10.1111/pan.12287. Epub 2013 Nov 15. PMID 24237879
- [Result] Yuen VM, Hui TW, Irwin MG, Yao TJ, Chan L, Wong GL, Shahnaz Hasan M, Shariffuddin II. A randomised comparison of two intranasal dexmedetomidine doses for premedication in children. Anaesthesia. 2012 Nov;67(11):1210-6. doi: 10.1111/j.1365-2044.2012.07309.x. Epub 2012 Sep 5. PMID 22950484
- [Derived] Sathyamoorthy M, Hamilton TB, Wilson G, Talluri R, Fawad L, Adamiak B, Wallace C, Borissova I, Heard C. Pre-medication before dental procedures: A randomized controlled study comparing intranasal dexmedetomidine with oral midazolam. Acta Anaesthesiol Scand. 2019 Oct;63(9):1162-1168. doi: 10.1111/aas.13425. Epub 2019 Jul 18. PMID 31318038

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midazolam | Dexmedetomidine
Started | 38 | 37
Completed | 37 | 36
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Dexmedetomidine | Total
Number analyzed (Participants) | 37 | 36 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 36 | 73
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.62 (2.3) | 8.0 (3.37) | 7.9 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 26 | 24 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 36 | 73

OUTCOME MEASURES:

1. Primary Outcome: University of Michigan Sedation Scale
Description: Level of sedation at separation from parents and at the time of mask induction will be measured on a scale of 0 to 4 (University of Michigan Sedation Scale)
  University of Michigan Sedation Scale:
  0 -Awake/Alert
  1 -Minimally Sedated: Tired/sleepy, appropriate response to verbal conversation and/or sounds.
  2- Moderately Sedated: Somnolent/sleeping, easily aroused with light tactile stimulation.
  3 - Deeply Sedated: Deep sleep, arousable only with significant physical stimulation.
  4 - Unarousable
  Moderately and Deeply sedated: Satisfactory Awake, minimally sedate, unarousable: Unsatisfactory
Time Frame: Day 0:Just before the patient will be brought to the operating room
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 37 | 36
Participants
  Satisfactory sedation on separation from parents | 15 | 25
  Unsatisfactory sedation on separation from parents | 22 | 11
  Satisfactory sedation on transfer to OR table | 12 | 22
  Unsatisfactory sedation on transfer to OR table | 25 | 14
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; A sample size of at least 33 patients in each group would detect at least 30% difference in proportion of children who achieve satisfactory sedation between the M and D groups at 0.05 level of significance and 80% power; Test type: Superiority or Other; p = 0.025, Chi-squared — Difference in proportions in satisfactory sedation on separation from parents and on induction between M and D groups (Primary Outcome variables)

2. Secondary Outcome: Acceptance of Mask Induction
Description: on a scale of 1 to 4
  1. excellent( cooperative)
  2. good( slight fear, easily calmed)
  3. fair ( moderate fear, not calmed with reassurance)
  4. Poor( agitated, terrified) 1 and 2 are considered satisfactory 3 and 4 are considered unsatisfactory
Time Frame: Day 0: At the time when anesthesia is induced
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 37 | 36
Participants
  Satisfactory mask induction | 35 | 29
  unsatisfactory mask induction | 2 | 7
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; Test type: Superiority or Other; p > 0.05, Chi-squared

3. Secondary Outcome: Wake up Behavior
Description: assessed in post anesthesia recovery unit after the procedure on a scale of 1o 4
  1. calm
  2. not calm but easily calmed
  3. moderately agitated or restless
  4. combative/disoriented 1 and 2 are considered satisfactory 3 and 4 are considered unsatisfactory
Time Frame: Day 0: At the end of surgery when the patient recovers from anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 37 | 36
Participants
  satisfactory wake up behavior | 37 | 35
  unsatisfactory wake up behavior | 0 | 1
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; Test type: Superiority or Other; p > 0.05, Chi-squared

4. Secondary Outcome: Presence of Amnesia to Mask Induction
Description: Yes or No (if the patient remembers mask induction)
Time Frame: Day 0: at the time of discharge of the patient from the recovery room
Population: 7 patients in the M group and 5 patients in D group had significant developmental delay and could not answer the question regarding memory of mask induction. Thus, only 61 were analyzed for this part
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 30 | 31
Participants
  memory of mask induction-yes | 6 | 5
  memory of mask induction-no | 24 | 26
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; Test type: Superiority or Other; p > 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: After premedication, patients will be continuously monitored including HR, BP, RR and SPO2 and documented every 15 min
Arm/Group | Midazolam | Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36
Other Adverse Events (participants affected / at risk) | 0/37 | 0/36

LIMITATIONS AND CAVEATS:
All the consecutive patients were screened for eligibility. Patients were not selected on the basis of need for premedication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes